CLINICAL TRIAL: NCT05547997
Title: The Efficacy of Cervical Lordosis Rehabilitation for Nerve Root Function and Pain in Cervical Spondylotic Radiculopathy: A Randomized Trial With 2-year Follow-up
Brief Title: The Efficacy of Cervical Lordosis Rehabilitation for Nerve Root Function and Pain in Cervical Spondylotic Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Professor-chair of Physiotherapy Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo-20-18-4
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Cervical Lordosis Rehabilitation
Keywords: Cervical spine; Lordosis; Dermatomal; Traction
MeSH Terms: conditions — Lordosis | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Parallel Assignment A prospective, double blinded, parallel-group, randomized clinical trial will be conducted at one of our university's research departments,
Who Masked: Outcomes Assessor
Masking Description: The assessor who will conduct the measurements will be blinded. Assessor blinding will be obtained through an independent research assistant not knowing the study design and not specifically involved in any aspect of the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- two way traction (Experimental): The study group will receive 3-point bending cervical extension traction following the protocol of Harrison et al. The duration of each session will starte at approximately three minutes and increased one minute per session until reaching the goal of 20 minutes per session
  Interventions: Other: Stretching exercises; Other: Two way traction
- traditional treatment (Active Comparator): Stretching exercises: Patients will perform the stretching program 3 times a week; with a single session taking about 10 minutes to perform.
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Other: Stretching exercises — Exercises will be performed in the following order: 1) stretching towards lateral flexion for the upper part of the trapezius; 2) ipsilateral flexion and rotation for the scalene; 3) and flexion for the extensor muscles. Each maneuver will be held for 30 seconds as this is an optimum time to not create alteration in the evoked protentional. Each stretch will be repeated 3 times
Other: Two way traction — During the traction, the head halter will be fixed posteriorly to cause slight distraction, retraction, and slight extension and at the same time a front anterior strap had weight will be applied over a pulley that allows transverse traction load to be applied to the apex of the participants cervical curve alteration. Weights will start at 15 lbs. (6.8 Kg) on the anterior strap and will increase over consecutive visits to patient tolerance or a maximum of 35 lbs. (15.9 Kg).
  Arms: two way traction

SUMMARY:
To test the hypothesis that improvement of cervical lordosis (CL) in cervical spondylotic radiculopathy (CSR) will improve clinical features in a population suffering from CSR. Thirty chronic lower CSR patients with CL < 25° will be included. Patients will be assigned randomly into two equal groups, study and control . Both groups will receive neck stretching and exercises and infrared; additionally the study group will receive cervical extension traction. Treatments will be applied 3 time per week for 10 weeks after which groups will be followed for 3-months and 2-years. Amplitude of dermatomal somatosensory evoked potentials (DSSEPS), Cervical lordosis, and pain scales (NRS) will be measured.

DETAILED DESCRIPTION:
Previous studies testing the effects of 3-point bending types of cervical traction, have not clarified exactly what impact the sagittal cervical curve correction has on nerve root function and pain responses associated with improving an abnormal cervical lordosis in cervical spondylotic patients. The present randomized controlled trial will be undertaken to investigate the neurophysiological and pain response outcomes of 3-point bending (2-way) traction compared to standard care in patient cases with lower cervical spine CSR, chronic pain, and with a verified hypo-lordosis of the cervical spine. The primary hypothesis of this study will be that cervical lordosis restoration will have short- and long-term effects on DSSEPs and pain outcomes in CSR patients.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral radiculopathy due to spondylotic changes of the lower cervical spine
* Absolute rotatory angle is less than 20°
* side to side amplitude differences of 50% or more in dermatomal somatosensory evoked potentials measurement

Exclusion Criteria:

* Central spinal canal stenosis
* Rheumatoid arthritis
* Vestibulobasilar insufficiency
* Osteoporosis
* Inability to tolerate the cervical extension position

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The Change in amplitude of dermatomal somatosensory evoked potentials | will be measured at four intervals ;before treatment, after 10 weeks of treatment, at follow up of 3 months and at follow up of 2 years
  In all dermatomes, two complete recording runs will be undertaken during each session, with averages of 250-1,200 cortical responses from scalp surface recording electrodes (C3'-C4' in a 10-20 electrode configuration) of the contralateral scalp to the C6, C7, and C8 dermatomes being stimulated

SECONDARY OUTCOMES:
The change in pain intensity | will be measured at four intervals ;before treatment, after 10 weeks of treatment, at follow up of 3 months and at follow up of 2 years
  Measurement of pain will be performed by using a visual analogue scale (VAS). The subjects will be asked about the perception of pain using a 10-cm line with 0 (no pain) on one end and 10 (worst pain) on the other. subjects will be asked to place a mark along the line to denote their level of pain

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Moustafa, Professor, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No